CLINICAL TRIAL: NCT03640689
Title: DEep VEin Lesion OPtimisation (DEVELOP) Trial: A Randomised, Assessor-blinded Feasibility Study of Iliac Vein Intervention for Venous Leg Ulcers
Brief Title: DEep VEin Lesion OPtimisation (DEVELOP) Trial
Acronym: Develop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Thomas Aherne, Principle Investigator Dr Thomas Aherne, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NUIreland1
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Venous Leg Ulcer
Keywords: Venous ulcer; Great saphenous incompetence; Iliac vein; Endovenous therapy
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Group (Experimental): Endovenous ablation + iliac US +/- iliac stenting
  Interventions: Device: Endovenous ablation + iliac US +/- iliac stenting
- Control Group (Active Comparator): Endovenous ablation of Great Saphenous Vein
  Interventions: Device: Endovenous ablation of Great Saphenous Vein

INTERVENTIONS:
Device: Endovenous ablation + iliac US +/- iliac stenting — Concomitant Ablation of the GSV with endovenous therapy with associated iliac vein interrogation and stenting if required
  Other Names: Graduated Compression Stockings; Iliac vein intravascular ultrasound; Iliac vein stenting
  Arms: Intervention Group
Device: Endovenous ablation of Great Saphenous Vein — Ablation of the Great Saphenous Vein and subsequent Graduated Compression
  Other Names: Graduated Compression Stockings
  Arms: Control Group

SUMMARY:
This is a prospective, single centre, randomised controlled, feasibility study recruiting patients with lower limb venous ulceration and Great Saphenous incompetence. Patients will be randomised to undergo either truncal ablation and compression therapy or truncal ablation, simultaneous iliac interrogation with intravascular ultrasound and stenting of significant (>50%) iliac vein lesions plus compression therapy. The primary endpoints will be ulcer healing and procedural safety. Secondary endpoints include time to healing, quality of life and clinical scores, ulcer recurrence rates and rates of post-thrombotic syndrome. Follow up will be over a five-year period. This feasibility study is designed to include 60 patients. Should it be practicable a total of 594 patients would be required to adequately power the study to definitively address ulcer-healing rates.

DETAILED DESCRIPTION:
The single main research question for this trial is as follows: in adult patients with venous ulceration and great saphenous vein incompetence; does iliac vein assessment with IVUS and stenting of significant occlusive disease in addition to superficial great saphenous venous ablation and compression compared to superficial venous ablation and compression alone offer improved ulcer healing rates at three months following treatment?

Primary Objective To determine whether superficial venous ablation plus early iliac vein interrogation plus endovascular stenting in the presence of significant occlusive disease results in improved venous ulcer healing compared to superficial venous ablation plus compression therapy alone.

Secondary Objectives

1. To determine the relative performance of duplex ultrasound compared to IVUS for the prediction of NIVLs 3. To determine the rate of primary or recurrent ulceration up to five years following intervention 4. To assess patient quality of life in the short and medium term following each mode of intervention

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients
* aged 18 and over
* ultrasound detected Great Saphenous Venous incompetence
* an associated primary or recurrent lower limb venous ulcer(s)

Exclusion Criteria:

* Ankle-brachial pressure index <0.8
* Previous inability to tolerate lower limb compression bandaging
* Inability to provide informed consent
* Previous lower limb arterial revascularisation procedure
* Contrast allergy
* Previous history of pelvic malignancy or pelvic radiotherapy
* Pregnancy
* Previous iliac vein intervention
* Previous superficial vein intervention
* Infection in previous 30 days
* Estimated glomerular filtration rate (eGFR) < 60 mls/kg/min
* Isolated short saphenous or perforator vein reflux only
* Leg ulcer of non-venous aetiology (as assessed by clinician)
* Unfit for endovascular intervention based on history and examination
* Any compression therapy within six-months
* Evidence of deep venous incompetence/thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Ulcer Healing - Proportion of ulcers healed | 3-months
  Proportion of ulcers healed
Iliac Vein Patency on duplex ultrasound | 6-months
  Patency of the iliac vein on duplex
Reintervention | 12-months
  Freedom from re-intervention

SECONDARY OUTCOMES:
Ulcer healing - Time to ulcer healing | In days
  Time to ulcer healing
Patient Quality of life using the Aberdeen Varicose Vein Questionnaire | 12-months
  Aberdeen Varicose Vein Questionnaire measured from 0(no effect)-100(severe effect). The higher the score the greater the negative impact on patient quality of life.
Recurrence - Ulcer recurrence | 12-months
  Ulcer recurrence

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Soalta Hospital Group, Galway
  - Univsersity Hospital Galway, Galway

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year for 5 years

REFERENCES:
- [Derived] Aherne TM, Keohane C, Mullins M, Zafar AS, Black SA, Tang TY, O'Sullivan GJ, Walsh SR. DEep VEin Lesion OPtimisation (DEVELOP) trial: protocol for a randomised, assessor-blinded feasibility trial of iliac vein intervention for venous leg ulcers. Pilot Feasibility Stud. 2021 Feb 4;7(1):42. doi: 10.1186/s40814-021-00779-2. PMID 33541436